CLINICAL TRIAL: NCT04615208
Title: A Touchless Tool to Screen for COVID-19 for Reopening Industries
Brief Title: Screening for COVID-19
Status: Withdrawn | Type: Observational
Why Stopped: due to complete lack of cooperation from Winnipeg Health authorities we were not able to recruit and enrolled any participant. We needed to recruit from visitors to testing stations and we were never allowed to do that.
Sponsor: University of Manitoba (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); ID Fusion Software, Inc. (Unknown); Function Four Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: B2020:070 (HS24165)
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: Covid19; screnning; touches
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: suspected of COVID-19 infection — suspected of COVID-19 infection

SUMMARY:
Canada is entering the important yet dangerous phase of the COVID-19 pandemic: the reopening of industry. As such, there is an urgent need for a quick and accurate screening tool to help ensure people re-entering the workplace are COVID-19 negative. This proposal offers an innovative, simple-to-implement and quick screening tool for this purpose. This study hypothesize that breathing sounds of a COVID-19 positive person would have different characteristics even if the person is asymptomatic. This study aim the development of an integrated diagnostic pattern recognition tool in the form of a smartphone app, using audio and temperature as inputs to identify COVID-19 positive individuals. The proposed digital technology will screen individuals as healthy or possibly COVID-19 positive. The latter group will then be recommended for further testing. The goal of the proposed app is to provide much more accurate early screening (currently only temperature is taken), and to reduce the burden of COVID-19 tests. This digital technology will be used and tested in Manitoba initially and later nationally in Canada, with the potential of being publicly available in the future.

To use the proposed screening tool, a smartphone is held within 1 cm of an individual's mouth and the individual instructed to take five deep breaths through the mouth. The individuals' breathing sounds will be recorded by the smartphone, while the participant's temperature will also be recorded by the heat camera. The app will first use its acoustic analysis to identify sounds as healthy or abnormal. If the outcome is abnormal, then a questionnaire will be provided, along with a further acoustic analysis to rule out other common comorbid conditions (e.g. chronic lung disease). Finally, based on the inputs, the diagnostic algorithm will decide if the individual should be referred for further testing or not. Since the proposed end product is a smartphone app, the two software partner companies will play a crucial role in the final integration and development.

DETAILED DESCRIPTION:
The goal of this project is to develop a digital technology including an interactive app on a dedicated smartphones to record, analyze and classify a person as likely COVID-19 positive or negative. The specific objectives are:

1. Develop an initial simple app to record breathing sounds, check the quality of sounds in real time, message and instruct if the sounds fail the quality check.
2. Recruit and collect breathing sounds of at least up to 200 individuals at one of the COVID-19 testing stations in Winnipeg.
3. Using data of 50 COVID-19 positive cases and 50 negative ones of the above collection as the training data, develop a breathing sounds analysis algorithm with high sensitivity and specificity for smartphones to classify the recorded breathings sounds as healthy or abnormal. Our current database allows for immediate detection of some underlying unrelated pathologies, which in the initial stages will be supported by the included questionnaire. This can be further enhanced at the end-product stage as each worker's history is built up and daily compared.
4. Develop a smart diagnostic algorithm for smartphones as an app using the above sound analysis outcome, the subject's temperature and answers to a few questions and screen for possibility of having Covid-19 in less than 30 seconds.
5. Evaluate the above diagnostic algorithm for the remaining collected data (100 subjects), and plan for the next phase of study as a triage in one of the city's hospitals.
6. Prepare the final market prototype of the technology and disseminate the results.

ELIGIBILITY:
Inclusion Criteria:

* Adults being tested for COVID-19 by swab fluid test
* Must have a smart phone and Internet access

Exclusion Criteria:

* age<18 years
* cognitively impaired
* having no access to a smart phone or Internet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults suspected of COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
being positive or negative on COVID-19 swab fluid test | one week
  Swab Fluid Test

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Moussavi, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Upon Ethics approval, we would like to share our recorded breathing sounds with public.